CLINICAL TRIAL: NCT06910462
Title: IPM Intervention for Family Child Care Home Directors
Brief Title: Reporting Back Pesticide Results to Family Child Care Home Directors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4000 317300 144257A 01; R01ES036261-01 (NIH)
Record Dates: First submitted 2025-03-13; First posted 2025-04-04 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Pesticide Exposure; Community-based; Family

STUDY DESIGN:
Intervention Model Description: The intervention will include resources about IPM practices and understanding the potential exposure to pesticides and health effects for family child care home staff and children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated Pest Management and Report Pesticide Exposure (Experimental): Provide integrated pest management (IPM) toolkit and results of dust sample identifying pesticide exposure.
  Interventions: Behavioral: Integrated pest management (IPM) practices

INTERVENTIONS:
Behavioral: Integrated pest management (IPM) practices — Provide IPM resources to family child care home directors along with information about their exposure to pesticides and use of pesticides to lower their health risks.
  Other Names: Reduce use of pesticides to lower health risks

SUMMARY:
Child Care Health Consultants will provide an integrated pest management (IPM) intervention for ~30 family child care home directors. The intervention will include an educational component, collecting carpet dust samples, reporting back the pesticides identified in the carpet, and 7-monthly consultations to identify ways to reduce their exposure to pesticides and lower their long term health risks.

DETAILED DESCRIPTION:
The 12-month IPM intervention study conducted in family child care homes will include baseline and post-intervention interviews with the family child care home director, surveys, environmental assessments, and carpet dust samples. The intervention will include an IPM educational meeting where the director will receive an IPM Toolkit and toolbox, learn about the health risks related to repeated pesticide use. Six monthly consultations will be provided to focus on the goals set by the director to increase their IPM practices, reduce their use of pesticides, and lower the health risks for the children in their care, themselves and their staff. Three months after baseline, study staff will share the results of the pesticides detected in the dust samples to individual family child care home directors using Digital Exposure Report-Back Interface (DERBI). Interviews throughout the study period will be conducted with the family child care home directors to explore their reactions to and understanding of results, health effects, decisions made, intention to change pest management strategies, and/or share the results with families and their community.

ELIGIBILITY:
Inclusion Criteria: Director of a family child care home with 5 or more children in San Joaquin, Stanislaus, Tulare, or Fresno County in California. Plan to stay open for at least 12 months.

Exclusion Criteria: Does not read or speak English or Spanish.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-04-02 (Estimated); Study Completion 2028-04-28 (Estimated)

PRIMARY OUTCOMES:
IPM practices | one year
  Increased IPM practices as identified on the standardized, observational IPM Checklist post-intervention.
Decrease Pesticide Use and Exposure in Family Child Care Home | one year
  Observational checklists will be used to identify the number of pesticide sprays in the family child care home. Carpet dust analyses conducted by Southwest Research Institute (SwRI) will identify the detection and concentration of pesticides in the carpet dust.

SECONDARY OUTCOMES:
Increased understanding of health risks associated with pesticide use | one year
  Qualitative analyses will be conducted on the director interviews to identify themes and knowledge of the health risks associated with pesticide use, alternative treatments, IPM approach to pest management comparing pre- versus post-intervention responses.

CONTACTS AND LOCATIONS:
Overall Officials: Abbey Alkon, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF School of Nursing, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hazard K, Alkon A, Gunier RB, Castorina R, Camann D, Quarderer S, Bradman A. Predictors of pesticide levels in carpet dust collected from child care centers in Northern California, USA. J Expo Sci Environ Epidemiol. 2024 Mar;34(2):229-240. doi: 10.1038/s41370-022-00516-8. PMID 36599924
- [Background] Alkon A, Gunier RB, Hazard K, Castorina R, Hoffman PD, Scott RP, Anderson KA, Bradman A. Preschool-Age Children's Pesticide Exposures in Child Care Centers and at Home in Northern California. J Pediatr Health Care. 2022 Jan-Feb;36(1):34-45. doi: 10.1016/j.pedhc.2021.09.004. Epub 2021 Oct 8. PMID 34629233
- [Background] Stephens M, Hazard K, Moser D, Cox D, Rose R, Alkon A. An Integrated Pest Management Intervention Improves Knowledge, Pest Control, and Practices in Family Child Care Homes. Int J Environ Res Public Health. 2017 Oct 26;14(11):1299. doi: 10.3390/ijerph14111299. PMID 29072618